CLINICAL TRIAL: NCT03965338
Title: Assessment of Brain Activity During Complex Fine Hand Movements: an fMRI Study
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nesil Coskunfirat, Associate Professor, Akdeniz University
Other Study IDs: 4508.24.12.2018; 4508 TSA-2019-4508 (Other: BAP-AKDENIZ UNIVERSITY)
Record Dates: First submitted 2019-05-20; First posted 2019-05-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Regional Anaesthesia; Functional Magnetic Resonance Imaging
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fMRI brain activity: screening
  Interventions: Diagnostic Test: fMRI

INTERVENTIONS:
Diagnostic Test: fMRI — Screening

SUMMARY:
Brain cortex controls movement but the influence of peripheral component of movement on the cortex is not known. Functional Magnetic Resonance Imaging(fMRI) studies in stroke and fantom limb patients investigate cortex areas activated during execution and imagination of complex hand movements. These studies aim to understand the mechanisms of the motor component of movement but the results are limited as there is no effector organ in fantom limb patients and the affecting organ is damaged in stroke patients. The investigators hypothesized that the areas of the cortex that is activated to remember, set-up and order to move can be isolated from the areas that are activated during the motor component of movement. To prove this hypothesis the investigators developed a model that investigate the brain activation areas during the patient try to execute and imagine doing a complex motor task (sequential opposition with the thumb to the other four fingers) with a peripherally blocked arm. Brain fMRI in 15 right-handed patients scheduled to undergo right-hand surgery with peripheral block anesthesia will be obtained before the surgery day and just before surgery after the block. Participants will be screened when executing the task (after the block they just attempt), during rest and during they imagine doing the task. Bilateral cortex activation areas will be compared when the right hand was intact and was peripherally blocked.

There are many unknowns in the relationship between the brain-peripheric organ during movement. The investigators hope that some of these mechanisms will be identified by the new model we used in our study. The final benefit will be to develop stroke therapies and new therapies for neuropathic pain which is closely related to motor function.

DETAILED DESCRIPTION:
In this study, the investigators aim to separate the cortex areas that are activated during one remember, set-up and plan and start doing a motor task from the areas that are activated during performing the motor component. The investigators hypothesized that these areas can be identified by screening areas with fMRI when participants are asked to perform a complex motor task with a hand that is completely blocked. The hypothesis is based on the fact that in a participant with a peripherally blocked arm the central component of the movement will not be affected and the activation areas that remember and plan to do a motor task can be separated from the areas that are activated when the effector organ is doing the motor task, in other words, the motor component of the task.

the investigators also aim to show;

1. If there is an ipsilateral cortex activity during a participant with a peripherally blocked arm try to execute a complex motor task. The investigators know that in centrally paralyzed hands there is ipsilateral activity and there is no argument if this is an adaptive response or it is present from the beginning of the motor paralysis due to the strength of the central event of the contralateral brain area.
2. If there is a difference between activation areas of the cortex during the imaginary of complex hand movements with the intact and peripherally blocked arms.

Adult patients (>18) that have been scheduled to have right-hand surgery with peripheral blockage of the arm will be evaluated for the study. The patients will be informed about all the details and the consequences of the study and patients who give written informed consent will be included in the study. Local ethics committee approval is obtained in 05.12.2018. the study will be continued until the planned 15 patients are recruited for the study.

Right-hand dominance of the patient will be confirmed by Edinburgh handedness inventory (Oldfield,1971) and scores will be recorded. In the end, the mean of the score will be obtained for the whole study population. medium-high degree right handedness will be required for inclusion to the study. The patients who do not give written informed consents, patients who use their left hand dominantly, patients who have a neurologic or psychiatric disease, the patients with hearing and visual loss, who have history of substance abuse or who had surgery in the previous 12 months, with a history of major systemic disease (ASA III and IV) , with history of drugs that alter neurologic activity, who are unable to stay at MR machine without sedation, who are accepted to have a surgery duration of more than 3 hours, and patients who have a motor deficit at their right hand that makes the performance of the motor task impossible will not be included to the study. before the MR scanning patients will have a neurologic examination to show any neurologic insult related to the pathology they will have the operation for.

All these examinations and evaluations will be made at most 10 days before surgery.

The participants will perform a given motor task of block sequence. Patients will touch the other digits by the thumb in a given order and sequence. At the same session patients, will be screened while imagining doing the same task. The orders to rest, imagine and perform the task will be given by an MRI compatible monitor- mirror set. Patients will practice the task of the experiment before the real screening sessions. The patients will be observed while in the magnet to see if they perform the task appropriately.

ELIGIBILITY:
Inclusion criteria: Patients

* >18 years
* have right-hand surgery with peripheral blockage of the arm
* who give written informed consent
* who are right-hand dominant Exclusion criteria: Patients
* who do not give written informed consents,
* use their left hand dominantly,
* have a neurologic or psychiatric disease,
* have hearing and visual loss,
* have a history of substance abuse
* have surgery in the previous 12 months,
* have major systemic disease(ASA III and IV),
* have history of drugs that alter neurologic activity,
* are unable to stay at MR machine without sedation,
* with an expected surgery duration of more than 3 hours,
* have a motor deficit at their right hand that makes the performance of the motor task impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to have right-hand surgery with peripheral blockage of the arm
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-04-12 (Actual)

PRIMARY OUTCOMES:
Compare the area of brain activation during the participant try to perform a motor task when the hand is blocked with area of brain activation when the hand actually perform the task by using fMRI | 1 year
  complex hand movement: sequential repetitive thumb to other four digit opposition with the right hand
Comparing brain activation areas while the participant imagine to perform a motor task when the hand is blocked with brain activation areas when the hand is intact, by fMRI | 1 year
  complex hand movement: sequential repetitive thumb to other four digit opposition with the right hand

SECONDARY OUTCOMES:
Comparing the area of ipsilateral cortex brain activity when the participant is intending to perform the complex motor task with the area while imagining doing the complex motor task when the arm is blocked by anesthesia. | 1 year
  complex hand movement: sequential repetitive thumb to other four digit opposition with the right hand

CONTACTS AND LOCATIONS:
Overall Officials: Utku A Senol, Prof., Principal Investigator — Akdeniz University Radiology Department
Locations (1):
- AkdenizU, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Bihan D, Karni A. Applications of magnetic resonance imaging to the study of human brain function. Curr Opin Neurobiol. 1995 Apr;5(2):231-7. doi: 10.1016/0959-4388(95)80031-x. PMID 7620312
- [Background] Ruffino C, Papaxanthis C, Lebon F. Neural plasticity during motor learning with motor imagery practice: Review and perspectives. Neuroscience. 2017 Jan 26;341:61-78. doi: 10.1016/j.neuroscience.2016.11.023. Epub 2016 Nov 25. PMID 27890831
- [Background] Osumi M, Sumitani M, Wake N, Sano Y, Ichinose A, Kumagaya S, Kuniyoshi Y, Morioka S. Structured movement representations of a phantom limb associated with phantom limb pain. Neurosci Lett. 2015 Sep 25;605:7-11. doi: 10.1016/j.neulet.2015.08.009. Epub 2015 Aug 10. PMID 26272300